CLINICAL TRIAL: NCT03809156
Title: Upfront Riociguat and Ambrisentan Combination Therapy for Pulmonary Arterial Hypertension: A Safety and Efficacy Pilot Study
Brief Title: Upfront Combination Pulmonary Arterial Hypertension Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-3056
Record Dates: First submitted 2019-01-09; First posted 2019-01-18 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combo Riociguat and Ambrisentan Therapy (Experimental): Riociguat Oral Product and Ambrisentan Oral Product to be given in combination to de novo (untreated) patients.
  Interventions: Drug: Riociguat Oral Product

INTERVENTIONS:
Drug: Riociguat Oral Product — Dual therapy of Riociguat and Ambrisentan at initiation of treatment.
  Other Names: Ambrisentan Oral Product

SUMMARY:
To evaluate the safety and efficacy of first-line combination therapy using riociguat with ambrisentan in patients with Pulmonary Arterial Hypertension (PAH).

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, exploratory study with patients followed for a period of one year. The treatment duration period in this study begins at the initiation of ambrisentan plus riociguat and will continue for 12 months. Patients will come to clinic for a visit at month 4 and 12. Assessments will include Right Heart Catheterization, 6 Minute walk test, cardiac MRI, questionnaires and nt-Pro-BNP.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study mandated procedure;
2. Males or females ≥ 18 years of age i. Women of childbearing potential must have a negative pre-treatment pregnancy test and must use reliable methods of contraception.

   ii. Women not of childbearing potential are defined as postmenopausal (i.e., amenorrhea for at least 1 year), or documented surgically or naturally sterile.
3. Patients with symptomatic Functional Class III PAH in the following categories:

   i. Idiopathic (IPAH) ii. Familial (FPAH) iii. Associated with connective tissue disease iv. Associated with drugs or toxins;
4. PAH diagnosed by right heart catheterization, defined as:

   i. Mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg ii. PVR > 3 mmHg/l/min (Wood units) or > 240 dyn sec cm-5 iii. Pulmonary capillary wedge pressure (PCWP) ≤ 15 mmHg;
5. 150 m ≤ 6 Minute Walk Test (6MWT) distance ≤ 480 m

Exclusion Criteria:

1. PAH associated with any other condition than those described in the inclusion criteria (patients with PAH associated with portal hypertension, HIV and CHD should not be included);
2. PAH associated with thyroid disorders, glycogen storage disease, Gaucher disease, hereditary hemorrhagic telangiectasia, hemoglobinopathies, myeloproliferative disorders and splenectomy;
3. Valvular disease with valvular lesions to be excluded by echocardiogram within 2 years prior to randomization (i.e., patients with tricuspid or pulmonary insufficiency secondary to PAH can be included);
4. Restrictive lung disease: total lung capacity (TLC) < 60% of normal predicted value;
5. Obstructive lung disease: forced expiratory volume/forced vital capacity (FEV1/FVC) < 0.5;
6. Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C;
7. Pregnancy or breast-feeding;
8. Systolic blood pressure < 95 mmHg;
9. Body weight < 40 kg;
10. Hemoglobin > 25% below the lower limit of the normal range;
11. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 1.5 times the upper limit of normal ranges;
12. Renal insufficiency as defined by creatinine clearance < 30 mL/min or on dialysis
13. Treatment with phosphodiesterase type 5 inhibitors, any prostanoid (excluding acute administration during a catheterization procedure to test vascular reactivity) or with any other PH specific medication;
14. Treatment or planned treatment with calcineurin-inhibitors (i.e., cyclosporine A and tacrolimus), CYP2C9 and CYP3A4 inhibitors (i.e., ketoconazole, fluconazole) within 1 week of study start;
15. Treatment or planned treatment with nitrate drugs, short acting nitrate-containing medications, alpha blockers or protease inhibitors (i.e., ritonavir);
16. Known hypersensitivity to ambrisentan, riociguat or any of their excipients;
17. Patients with any contraindication to riociguat treatment or ERA treatment
18. Patients with syncope, a rapid rate of symptom progression or with high or rising nt-BNP levels in the judgment of the investigators
19. Any contraindications specified in the product monographs of either ambrisentan or riociguat, including:

1. Patients at increased risk of hypotension with concomitant or underlying conditions such as coronary artery disease, hypovolemia, severe left ventricular outflow obstruction or autonomic dysfunction; patients with resting hypotension 2. Patients with history of serious hemoptysis or patients who have previously undergone bronchial arterial embolization 20. Patients with pulmonary veno-occlusive disease 21. Ongoing participation in any interventional clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-04-26 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Vascular resistance | 4 and 12 months
  Change from baseline to month 4 and month 12 in pulmonary vascular resistance (PVR) as assessed by Right Heart Catheterization.

SECONDARY OUTCOMES:
Hemodynamic Variables | 4 and 12 months
  Change in hemodynamic variables (mPAP, RAP, CI) from baseline to month 4 and month 12 as assessed by Right Heart Catheterization.
Echocardiographic parameters | 4 and 12 months
  Change in echocardiographic parameters (TAPSE, RV strain, Tei index, Left ventricular Eccentricity index, RV:LV area ratio) as assessed by Echocardiogram.
RV function | 4 and 12 months
  Change from baseline to month 4 in RV function as assessed by cardiac MRI.
NT-PRo-BNP | 4 and 12 Months
  Change from baseline NT-PRo-BNP value from baseline to month 4 and month 12
Exercise capacity | 4 and 12 months
  Change from baseline to month 4 and month 12 in exercise capacity assessed by the 6 minute walk test
Dyspnea | 4 and 12 months
  Change from baseline to month 4 and month 12 in dyspnea as assessed by study questionnaire.
Quality of Life Assessment | 4 and 12 months
  Change from baseline to month 4 and month 12 in quality of life as assessed by study questionnaire.
Functional Class | 4 and 12 months
  Change from baseline to month 4 and month 12 in functional class as assessed by study questionnaire.
Survival | 12 months
  Survival at 12 months
Clinical worsening | 12 months
  Time to clinical worsening over 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Naushad Hirani, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Peter Lougheed Center, Calgary, Alberta
  - Vancouver General Hospital, The Lung Centre, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No